CLINICAL TRIAL: NCT00010114
Title: Gene Expression Profiling of Infant Embryonal Central Nervous System Tumors by Microarray Gene Chip Analysis: Angiogenesis, Invasion and Metastasis
Brief Title: Genetic Study of Newly Diagnosed Central Nervous System Tumors in Young Children
Status: Completed | Type: Observational
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett, Executive Director Operations and Biostatistics Center, Pediatric Brain Tumor Consortium
Other Study IDs: CDR0000068446; PBTC-N04
Record Dates: First submitted 2001-02-02; First posted 2003-06-06 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Central Nervous System Embryonal Neoplasm
Keywords: childhood central nervous system germ cell tumor; childhood choroid plexus tumor; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma; newly diagnosed childhood ependymoma
MeSH Terms: conditions — Choroid Plexus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly diagnosed embryonal tumors: The participants in this study are infants (< 3 years of age) with newly diagnosed medulloblastoma, primitive neuroectodermal tumor, or other embryonal tumor, atypical teratoid/rhabdoid tumor, intracranial germ cell tumor, or choroid plexus carcinoma who have received no prior therapy with the exception of steroids and have consented to allow research studies on banked tissue specimens

SUMMARY:
RATIONALE: Genetic studies may help in understanding the genetic processes involved in the development of some types of cancer.

PURPOSE: Genetic study to learn more about genes involved in the development of central nervous system tumors in young children.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify known genes that have significantly different levels of expression, using microarray gene chip analysis, in infants with newly diagnosed metastatic vs non-metastatic embryonal central nervous system tumors.
* Determine the protein expression of genes identified by microarray analysis that are involved in cellular functions that regulate angiogenesis, invasion, or metastasis in this patient population.
* Determine the quantity of gene expression of the confirmed translationally expressed genes using semi-quantitative polymerase chain reaction.

OUTLINE: This is a multicenter study.

Tumor samples are analyzed using microarray gene chip analysis. Differentially expressed genes are evaluated for protein expression by standard immunohistochemistry and/or Western blot analysis, and gene expression is further quantified by semi-quantitative polymerase chain reaction.

PROJECTED ACCRUAL: Approximately 80-100 patients (20-25 with metastatic disease and 60-75 with non-metastatic disease) will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed, newly diagnosed, primary intracranial embryonal central nervous system tumor

  * Medulloblastoma
  * Primitive neuroectodermal tumor
  * Medulloepithelioma
  * Ependymoblastoma
  * Neuroblastoma
  * Pineoblastoma
  * Atypical teratoid/rhabdoid tumor
  * Intracranial germ cell tumor
  * Choroid plexus carcinoma
  * M positive ependymoma
* Potential enrollment on PBTC-001 therapeutic protocol

PATIENT CHARACTERISTICS:

Age:

* Under 3

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior steroids allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Other:

* No concurrent investigational agents

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The participants in this study are infants (< 3 years of age) with newly diagnosed medulloblastoma, primitive neuroectodermal tumor, or other embryonal tumor, atypical teratoid/rhabdoid tumor, intracranial germ cell tumor, or choroid plexus carcinoma who have received no prior therapy with the exception of steroids and have consented to allow research studies on banked tissue specimens
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2001-03; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Genes that are expressed in metastatic vs. non-metastatic tumors | Prior to therapy

SECONDARY OUTCOMES:
Protein expression of genes found to be expressed | Prior to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Tobey MacDonald, MD, Study Chair — Children's National Research Institute
Locations (9):
- United States (9):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington